CLINICAL TRIAL: NCT05736458
Title: Network Control and Functional Context: Mechanisms for TMS Response
Brief Title: Network Control TMS fMRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because our funding agency, the NIH, did not grant a no-cost extension to meet our recruitment goals.
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 830174; RF1MH116920 (NIH)
Record Dates: First submitted 2023-01-19; First posted 2023-02-21 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder; Working Memory
Keywords: TMS; memory; ADHD; healthy; MRI; ADD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All healthy participants will have TMS administered to both their high and low regional controllability targets, but the order is randomized and counterbalanced.
  ADHD participants will have TMS administered to only their high regional controllability target.
Who Masked: Participant
Masking Description: This study will use a single-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- High regional controllability TMS target in non-symptomatic participants (Experimental): We will administer TMS to an individualized target of high regional controllability while non-symptomatic participant completes a working memory task inside the MRI scanner.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Procedure: High controllability TMS target
- Low controllability TMS target in non-symptomatic participants (Active Comparator): We will administer TMS to an individualized target of low regional controllability while non-symptomatic participant completes a working memory task inside the MRI scanner.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- High regional controllability TMS target in ADHD participants (Experimental): We will administer TMS to an individualized target of high regional controllability while patient completes a working memory task inside the MRI scanner.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Procedure: High controllability TMS target

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication.
Procedure: High controllability TMS target — Administer TMS to a brain regions with high regional controllability while the subject engages in a working memory task.
  Arms: High regional controllability TMS target in ADHD participants; High regional controllability TMS target in non-symptomatic participants

SUMMARY:
This study uses different types of functional magnetic resonance imagining (fMRI) to generate individual transcranial magnetic stimulation (TMS) targets. During the TMS/fMRI imagining sessions, the investigators stimulate a target of either high or low regional controllability during a working memory task to investigate network responses and the impact of TMS on behavior.

DETAILED DESCRIPTION:
This study involves up to 4 visits for patients with Attention Deficit Hyperactivity Disorder (ADHD) and 5 visits for non-symptomatic subjects.

Visit 1 has both remote and in-person procedures. The remote part of visit 1 will consist of a consenting and extended screening visit. The in-person procedures of visit 1 will be scheduled for the same day as visit 2. Before visit 2, the investigators will demonstrate TMS to make sure participants can tolerate the stimulation.

Visit 2 consists of an hour-long baseline MRI Scan along with an assessment session. The baseline MRI scan is used to find individualized TMS targets. The assessment session of visit 2 will be done over a video call. During the video call, the investigators will have the participant complete some computerized tasks and assessments.

Visit 3 will be a 1-hour long TMS/fMRI session, where the participant will complete a working memory task twice while single pulse TMS is being delivered. In between the 2 rounds of the working memory task, the participant will receive 4 minutes of repetitive stimulation.

Non-symptomatic subjects will have a fourth visit that mirrors visit 3.

Visit 5 or Visit 4 for ADHD participants, will take place if behavioral task is available, otherwise study participation will be considered complete. During the optional visit, participants may complete behavioral tasks during an MRI scan. No TMS will be administered during the final visit.

Participants will receive the compensation at the end of their participation. Payment may be given earlier if the participant withdraws from the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-28 years old
* Right-handed
* No history of schizophrenia or bipolar disorder
* No history of neurological illness
* Healthy participants: no history of any mental illness
* ADD/ADHD Participants; Diagnosed with ADD/ADHD
* ADD/ADHD: Ability to refrain from stimulant medication within 24 hours of study sessions
* For participants reporting daily use of more than 400mg caffeine/ day: willing to lower down to this level at least 1 week prior to screening visit and maintain throughout study visits

Exclusion Criteria:

* Unable to have an MRI scan
* Unable to receive or tolerate TMS
* Pregnant, nursing, or trying to become pregnant (self-attestation alone)
* History of stoke, epilepsy, or brain scarring
* Healthy participants: psychoactive medication use
* Healthy participants: first degree relative with psychosis
* ADHD participants: inability to refrain from stimulant medication within 23 hours of study sessions
* Active suicidality or current suicidal risk as determined by the investigator
* Any medication that interferes with fMRI recordings as per PI discretion
* Otherwise determined by investigator to be unfit for study

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 68 participants screened for the study, 45 were enrolled and 23 did not start study procedures (13 screen failed, 4 withdrew from participation, and 6 lost to follow-up)
Groups:
- Non-symptomatic Participants High Modal Controllability First, Then Low Modal Controllability Target: Non-symptomatic participants will complete 2 TMS/fMRI visits, first receiving TMS to a high modal controllability target then the alternate low modal controllability target for the second TMS/fMRI.
  We will administer TMS to an individualized target of high & low modal controllability while asymptomatic participant completes a working memory task inside the MRI scanner.
  Transcranial Magnetic Stimulation (TMS): Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication.
  High controllability TMS target: Administer TMS to a brain regions with high modal controllability while the subject engages in a working memory task.
- Non-symptomatic Participants Low Modal Controllability First, Then High Modal Controllability Target: Non-symptomatic participants will complete 2 TMS/fMRI visits, first receiving TMS to a low modal controllability target then the alternate high modal controllability target for the second TMS/fMRI.
  We will administer TMS to an individualized target of high & low modal controllability while asymptomatic participant completes a working memory task inside the MRI scanner.
  Transcranial Magnetic Stimulation (TMS): Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication.
  High controllability TMS target: Administer TMS to a brain regions with high modal controllability while the subject engages in a working memory task.
- High Modal Controllability TMS Target in ADHD Participants: We will administer TMS to an individualized target of high regional controllability while patient completes a working memory task inside the MRI scanner.
  Transcranial Magnetic Stimulation (TMS): Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication.
  High controllability TMS target: Administer TMS to a brain regions with high modal controllability while the subject engages in a working memory task.
Period: Baseline MRI and Assessments
Arm/Group | Non-symptomatic Participants High Modal Controllability First, Then Low Modal Controllability Target | Non-symptomatic Participants Low Modal Controllability First, Then High Modal Controllability Target | High Modal Controllability TMS Target in ADHD Participants
Started | 13 | 13 | 19
Completed | 11 | 13 | 15
Not Completed | 2 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: TMS/fMRI #1
Arm/Group | Non-symptomatic Participants High Modal Controllability First, Then Low Modal Controllability Target | Non-symptomatic Participants Low Modal Controllability First, Then High Modal Controllability Target | High Modal Controllability TMS Target in ADHD Participants
Started | 11 | 13 | 15
Completed | 11 | 13 | 13
Not Completed | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 2
Period: Washout (at Least 7 Days)
Arm/Group | Non-symptomatic Participants High Modal Controllability First, Then Low Modal Controllability Target | Non-symptomatic Participants Low Modal Controllability First, Then High Modal Controllability Target | High Modal Controllability TMS Target in ADHD Participants
Started | 11 | 13 | 0 (ADHD Participants only complete TMS/fMRI #1)
Completed | 11 | 12 | 0
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: TMS/fMRI #2 (Only for Non-symptomatic)
Arm/Group | Non-symptomatic Participants High Modal Controllability First, Then Low Modal Controllability Target | Non-symptomatic Participants Low Modal Controllability First, Then High Modal Controllability Target | High Modal Controllability TMS Target in ADHD Participants
Started | 11 | 12 | 0 (ADHD Participants only complete TMS/fMRI #1)
Completed | 11 | 12 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-symptomatic Participants: Non-symptomatic participants or those without any psychiatric history complete two visits involving functional MRI (fMRI) and TMS. Each visit targets a specific brain controllability region, with one visit focusing on a high controllability region and the other on a low controllability region.
- ADHD Participants: Participants diagnosed with ADHD or ADD complete one visit involving functional MRI (fMRI) and TMS. This visit focuses exclusively on a high controllability brain region.
- Total: Total of all reporting groups
Arm/Group | Non-symptomatic Participants | ADHD Participants | Total
Number analyzed (Participants) | 26 | 19 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.96 (2.89) | 22.68 (1.86) | 22.84 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 23 | 17 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 15 | 13 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 19 | 45
E-SWAN ADHD scale [Mean (Standard Deviation); unit: units on a scale] — The Extended Strengths and Weaknesses of Attention-Deficit/Hyperactivity Symptoms and Normal Behavior Scale (E-SWAN) was administered via survey on their baseline MRI to assess ADHD symptoms. This scale includes 18 items rated from -3 (far below average) to 3 (far above average), divided into two subscales: Inattention and Hyperactivity/Impulsivity. Average scores for each subscale are used to interpret results. An average score above 0.745 on a subscale indicates presence of ADHD symptoms, with higher scores reflecting more severe symptoms and negative scores suggesting fewer or no symptoms.
  units on a scale
    Inattentive ADHD Subscale | -1.310 (0.730) | 0.750 (0.810) | -0.440 (1.28)
    Hyperactive/Impulsive ADHD Subscale | -1.300 (0.940) | 0.550 (0.840) | -0.520 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Single TMS Pulses to a High vs. Low Regional Controllability Target on Working Memory Task Performance
Description: Control participants complete two visits in which they undergo functional MRI interleaved with TMS targeting a specific controllability region. Each visit involves administering single pulses of TMS while participants perform a working memory task (N-back), followed by a brief round of repetitive TMS (rTMS), and concluding with another set of single pulses while completing the N-back task. The targeted brain region is counterbalanced across visits, with one visit stimulating a high regional controllability target and the other stimulating a low regional controllability target.
  The effect of single-pulse TMS on N-back task performance will be assessed before rTMS administration using percent accuracy scores. Percent accuracy reflects the percentage of correct trials out of the total Nback trials, with higher scores indicating better task performance.
Time Frame: Up to 3 weeks
Population: Of the 23 participants who completed all study procedures, 2 participants were unusable for this analysis.
Measure: Mean (95% Confidence Interval); unit: percentage of accuracy
Groups:
- TMS to a High Controllability Target in Non-Symptomatic Participants: Non-symptomatic participants undergoing functional MRI (fMRI) interleaved with TMS to a high controllability region.
- TMS to a Low Controllability Target in Non-Symptomatic Participants: Non-symptomatic participants undergoing functional MRI (fMRI) interleaved with TMS to a low controllability region.
Arm/Group | TMS to a High Controllability Target in Non-Symptomatic Participants | TMS to a Low Controllability Target in Non-Symptomatic Participants
Number analyzed (Participants) | 21 | 22
percentage of accuracy | 79.71 [69.96 to 89.45] | 78.39 [70.45 to 86.33]
Statistical Analysis 1: Comparison: TMS to a High Controllability Target in Non-Symptomatic Participants vs TMS to a Low Controllability Target in Non-Symptomatic Participants; Of the 23 participants who completed all study procedures, 2 participant's data was unusable for this analysis. Statistics are from paired 2 tailed t-test comparing pre-rTMS 2-back percent accuracy scores for participant's high and low controllability target; Test type: Superiority; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = 0.45

2. Primary Outcome: Effect of rTMS on Working Memory Task Performance
Description: Control participants complete two visits with functional MRI interleaved with TMS targeting a specific controllability region. Each visit includes single pulses of TMS during a working memory task (N-back), followed by a brief round of repetitive TMS (rTMS), and concluding with another set of single pulses while performing the N-back task. The targeted controllability region is counterbalanced, with one visit stimulating a high controllability target and the other a low controllability target.
  The effect of rTMS on N-back task performance will be assessed by comparing participants' percent accuracy scores before (pre-rTMS) and after (post-rTMS) rTMS. Percent accuracy, indicating the percentage of correct trials, will be analyzed for both high and low regional controllability targets across the visits.
Time Frame: Pre- and post-TMS at visits 3 (approximately day 7) and 4 (approximately day 14)
Population: Of the 23 participants who completed all study procedures, 2 participant's data was unusable for this analysis for the percent change comparison and high controllability group. Only 1 participant was unusable for the low controllability group.
Measure: Mean (95% Confidence Interval); unit: percentage accuracy
Arm/Group | TMS to a High Controllability Target in Non-Symptomatic Participants | TMS to a Low Controllability Target in Non-Symptomatic Participants
Number analyzed (Participants) | 21 | 22
percentage accuracy
  Nback results Pre-rTMS | 79.71 [69.96 to 89.45] | 78.39 [70.45 to 86.33]
  Nback results Post-rTMS | 81.65 [73.40 to 89.90] | 84.75 [77.57 to 91.93]
Statistical Analysis 1: Comparison: TMS to a High Controllability Target in Non-Symptomatic Participants; Statistics are from 2-tailed t-test comparing pre-rTMS to post-rTMS 2-back accuracy scores for a high controllability TMS target. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p = 0.43, t-test, 2 sided; df = 19; Mean Difference (Final Values) = 1.94
Statistical Analysis 2: Comparison: TMS to a Low Controllability Target in Non-Symptomatic Participants; Statistics are from 2-tailed t-test comparing pre-rTMS and post-rTMS 2-back percent accuracy scores for a low controllability TMS target. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p < 0.04, t-test, 2 sided; df = 20; Mean Difference (Final Values) = 6.36

3. Secondary Outcome: Effect of rTMS on Working Memory Performance in Participants With ADHD
Description: Participants with ADHD complete a single visit where they undergo functional MRI interleaved with TMS to a high controllability region. During the visit, participants receive single pulses of TMS while performing the working memory task (N-back), followed by a brief round of repetitive TMS (rTMS), and concluding with another set of single pulses while completing the N-back task.
  The effect of rTMS on N-back task performance is assessed by comparing participants' percent accuracy scores before (pre-rTMS) and after (post-rTMS) rTMS. Percent accuracy reflects the percentage of correct trials out of the total number of N-back trials, with higher percent accuracy indicating better performance.
Time Frame: Pre- and post-TMS at visit 3 (approximately day 7)
Population: Of the 13 participants with ADHD that completed the study, 1 participant's data was unusable for this analysis.
Measure: Mean (95% Confidence Interval); unit: percentage of accuracy
Groups:
- TMS to a High Controllability Target in Participants With ADHD: Participants diagnosed with ADHD/ADD complete one visit involving functional MRI (fMRI) and TMS targeting a high controllability region. During this visit, participants receive single pulses of TMS while performing a working memory task (N-back), followed by repetitive TMS (rTMS), and then another round of single pulses while completing the N-back task. Unlike non-symptomatic subjects, ADHD participants do not have a separate visit with TMS to a low controllability target.
Arm/Group | TMS to a High Controllability Target in Participants With ADHD
Number analyzed (Participants) | 12
percentage of accuracy
  Nback results Pre-rTMS | 69.64 [57.21 to 82.08]
  Nback results Post-rTMS | 81.18 [70.12 to 92.25]
Statistical Analysis 1: Comparison: TMS to a High Controllability Target in Participants With ADHD; Statistics are from 2-tailed paired t-test comparing 2-back accuracy score before and after rTMS to a high controllability target. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p < 0.05, t-test, 2 sided; df = 11; Mean Difference (Final Values) = 11.54

4. Primary Outcome: Effect of rTMS to High vs. Low Controllability Target on Working Memory Task Performance
Description: Control participants complete two visits where they undergo functional MRI interleaved with TMS targeting specific brain controllability regions. Each visit includes single pulses of TMS during a working memory task (N-back), followed by a brief round of repetitive TMS (rTMS), and concluding with another set of single pulses while performing the N-back task. The targeted brain region is counterbalanced across visits, with one visit stimulating a high controllability target and the other a low controllability target.
  In order to compare the effect of rTMS to high versus low controllability targets on working memory performance, we will assess the change in N-back task percent accuracy scores before (pre-rTMS) and after (post-rTMS) rTMS to both regions. A greater percent change (positive value) means improved task performance following rTMS.
Time Frame: Up to 3 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage accuracy change
Arm/Group | TMS to a High Controllability Target in Non-Symptomatic Participants | TMS to a Low Controllability Target in Non-Symptomatic Participants
Number analyzed (Participants) | 21 | 22
percentage accuracy change | 1.94 [-3.11 to 6.99] | 6.36 [0.57 to 12.16]
Statistical Analysis 1: Comparison: TMS to a High Controllability Target in Non-Symptomatic Participants vs TMS to a Low Controllability Target in Non-Symptomatic Participants; Statistics are from paired 2 tailed t-test comparing 2-back percent changes (Post-rTMS - pre-rTMS) scores for participant's high and low controllability target. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p = 0.27, t-test, 2 sided; df = 19; Mean Difference (Net) = -4.42

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study enrollment until study completion (up to 3 weeks).
Groups:
- High & Low Modal Controllability TMS Target in Non-symptomatic Participants: Non-symptomatic participants will complete 2 TMS/fMRI visits with alternate targets for a high and low modal controllability target.
  We will administer TMS to an individualized target of high & low modal controllability while asymptomatic participant completes a working memory task inside the MRI scanner.
  Transcranial Magnetic Stimulation (TMS): Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication.
  High controllability TMS target: Administer TMS to a brain regions with high modal controllability while the subject engages in a working memory task.
Arm/Group | High & Low Modal Controllability TMS Target in Non-symptomatic Participants | High Modal Controllability TMS Target in ADHD Participants
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/19
Other Adverse Events (participants affected / at risk) | 0/26 | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 4.44% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High & Low Modal Controllability TMS Target in Non-symptomatic Participants (N=26) | High Modal Controllability TMS Target in ADHD Participants (N=19)
Headache, dizziness, and nausea (General disorders) | 0 (0) | 1 (1) — Subject reported headache, dizziness, and nausea during TMS/fMRI. TMS was stopped and subject withdrew from study.
Minor Discomfort (General disorders) | 0 (0) | 1 (1) — Subject reported weird feeling in ear while receiving rTMS inside the MRI.

LIMITATIONS AND CAVEATS:
Enrollment goals were not completed due to delays resulting from COVID and not being granted a second no-cost extension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT05736458/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05736458/ICF_001.pdf